CLINICAL TRIAL: NCT01940367
Title: Percutaneous Tibial Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Overactive Bladder: A Randomized Trial
Brief Title: Electrical Nerve Stimulation for Overactive Bladder a Comparison of Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: International Urogynecological Association (Other); Section on Women's Health (Grant) (Unknown)
Responsible Party: Principal Investigator, Shannon Lamb, Physician, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 385408-2
Record Dates: First submitted 2013-08-13; First posted 2013-09-12 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Overactive Bladder; Urge Urinary Incontinence
Keywords: Overactive Bladder; TENS; PTNS; Electrical Nerve Stimulation; Urge Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTNS Arm (Active Comparator): Subjects randomized to the PTNS arm will undergo PTNS treatment once weekly for 30 minutes for 12 weeks total. If at 12 weeks they are considered to have a positive response to therapy, they will continue maintenance therapy in a tapered fashion: subjects will come in every 2 weeks for the next 8 weeks for 30 minute treatments (4 visits total), then every 3-4 weeks for 30 minute treatments for the remaining 32 weeks of the year (8-10 visits).
  Interventions: Device: PTNS (Percutaneous Tibial Nerve Stimulation
- TENS Arm (Active Comparator): Subjects randomized to the TENS arm of the study will begin therapy after their baseline evaluation is complete. They will be issued a home TENS device (EMPI TENS Select) and will administer self-treatment daily for 2 hours per day (1 hour in the morning and 1 hour in the evening) for a total of 12 weeks. If they are considered to have a positive response with TENS treatment, subjects will continue by weaning use over a three-month time period. They will begin with 3 x per week for 1 month, then 2 x per week for 1 month, then 1 x per week for 1 month, all at 2 hours per day.
  Interventions: Device: TENS (Transcutaneous Electrical Nerve Stimulation)

INTERVENTIONS:
Device: PTNS (Percutaneous Tibial Nerve Stimulation — PTNS therapy is performed as follows; the subject sits in a frog leg position in a chair. The area where the needle will be placed is cleaned with an alcohol swab. A 34 gauge needle (equivalent to an acupuncture needle) is inserted percutaneously approximately 5 cm cephalad to the medial malleolus of the right or left ankle (subject choice) at a 60 degree angle. A surface electrode is placed on the medial aspect of the ipsilateral calcaneous. The needle and electrode are connected to a low voltage (9 V) electrical stimulator (Urgent PC). Stimulation current with a fixed frequency of 20 Hz and a pulse width of 200 msec is increased until flexion of the big toe or fanning of all toes becomes visible, or until the subject reports a tingling sensation across the heel or bottom of the foot. The current is then set to the highest level tolerable to the subject (0-10 mA) and the subject undergoes therapy for 30 minutes.
  Other Names: Urgent ® PC Neuromodulation System
  Arms: PTNS Arm
Device: TENS (Transcutaneous Electrical Nerve Stimulation) — TENS therapy will be administered as follows:
  * Surface electrodes, 2" x 2" in diameter, will be placed over sacral foramen S2-4, bilaterally, using 2 channels (4 electrodes total) - Approximate locations are over posterior superior iliac spine and inferior lateral angle of sacrum. Sticker electrodes for the duration of the study will be issued to subjects. They are adhesive and can be re-used for up to 3-4 weeks with proper skin care and electrode care.
  * The electrodes will be connected to the TENS (Transcutaneous Electrical Nerve Stimulation) device and the following settings will be pre-set:
    * Mode: Burst
    * Cycle: 10 seconds
    * Frequency: 10 Hz
    * Pulse Width: 250 µs
    * Intensity: to subject comfort level
  Other Names: EMPI TENS Select
  Arms: TENS Arm

SUMMARY:
The purpose of this study is to determine whether transcutaneous sacral nerve stimulation (TENS SNS) versus percutaneous tibial nerve stimulation (PTNS) is a more effective therapeutic option for subjects with idiopathic overactive bladder (OAB) who have failed conventional therapy. Our primary hypothesis is that TENS therapy is a more effective treatment option due to ease of use and improved subject compliance with this form of therapy.

DETAILED DESCRIPTION:
To compare the long-term efficacy, subject compliance, and subject satisfaction of percutaneous tibial nerve stimulation (PTNS) therapy versus transcutaneous electrical sacral nerve stimulation (TENS) for the treatment of subjects with idiopathic overactive bladder. Previous short-term studies suggest that these therapies have equal efficacy in improving OAB symptoms, but we hypothesize that long-term efficacy and success is actually higher in the TENS group due to ease of use, since subjects can self-administer this therapy. Secondary goals are to evaluate subject quality of life improvement scores, bladder diary scores (change in the frequency of urination), and changes in urodynamic studies while undergoing these therapies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age >18 years
* Predominant complaint urge urinary incontinence (3 or more episodes per week) OR overactive bladder (8 or more voids per day, and/or 2 or more voids per night)
* Failed trial of conservative therapy (bladder training, fluid modification, diet modification, caffeine restriction, pelvic floor training)
* Failed trial of anticholinergic either due to inability to take the medication, adverse reaction to medication, or no improvement on medication
* Willing and mentally competent to participate in study
* Willing to complete study questionnaires
* No contraindications to undergoing PTNS or TENS therapy

Exclusion Criteria:

* Age < 18 years
* Presence of urinary fistula
* Male. (Males will be excluded because of the different etiology of overactive bladder for males which is primarily caused by prostate problems for men versus the primarily idiopathic cause in women).
* Recurrent or current urinary tract infection (5 or more infections in the last 12 months)
* Bladder stones
* Bladder cancer or suspected bladder cancer
* Hematuria
* Pregnancy or planning to become pregnant during the study (urine pregnancy test will be administered to those who are premenopausal and who have not had a hysterectomy)
* Central or peripheral neurologic disorders such as Multiple Sclerosis, Parkinson's disease, spina bifida, or other spinal cord lesion
* Metal implants such as pacemaker, implantable defibrillator, or metal implants where PTNS or TENS device needs to be placed (sacrum or ankle/leg).
* Uncontrolled diabetes
* Diabetes with peripheral nerve involvement
* On anticoagulants
* Current use of anticholinergics or use within the last 4 weeks
* Current use of botox bladder injections or bladder botox injection within the last year
* Current use of interstim therapy or currently implanted interstim device or leads
* Bladder outlet obstruction
* Urinary retention or gastric retention
* Painful Bladder Syndrome/Interstitial Cystitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Percutaneous Tibial Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Overactive Bladder: A Randomized Trial | 2 years
  The primary response variable is 'success' at 1 year, defined as a 50% or more reduction in the total number of incontinence episodes, or a 25% or more reduction in number of daily or nightly voids AND that the patient continues to use the therapy at one year. Therefore primary response is: 50% reduction in incontinence, OR 25% reduction in nightly voids AND continued use of therapy at one year.

SECONDARY OUTCOMES:
Percutaneous Tibial Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Overactive Bladder: A Randomized Trial | 2 years
  Participant compliance defined as 75% adherence to the recommended use for each device.
Percutaneous Tibial Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Overactive Bladder: A Randomized Trial | 2 Years
  Changes in the OAB-q (Overactive Bladder Questionnaire), the PFDI (Pelvic Floor Distress Inventory), and the FSFI (Female Sexual Function Index)
Percutaneous Tibial Nerve Stimulation vs. Transcutaneous Electrical Nerve Stimulation for Overactive Bladder: A Randomized Trial | 2 Years
  Changes in urodynamic studies (i.e. bladder capacity, uroflow rate, post-void residual).

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McVearry, DPT, WCS, Principal Investigator — Walter Reed National Military Medical Center
Locations (3):
- United States (3):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Portsmouth Naval Hospital, Portsmouth, Virginia